CLINICAL TRIAL: NCT00868101
Title: The Use of Remote Ischemic Preconditioning Applied in Child the Day Before Open Heart Surgery With Extracorporeal Circulation to Correct Congenital Heart Diseases (the Second Window Effect)
Brief Title: The Effect of Remote Ischemic Preconditioning Applied in Children the Day Before Open Heart Surgery
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Marcos Alves Pavione, mester, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MAP01
Record Dates: First submitted 2009-03-23; First posted 2009-03-24 (Estimated); Results first posted 2012-01-09 (Estimated); Last update posted 2012-01-09 (Estimated); Status verified 2011-12

CONDITIONS: Congenital Heart Disease
Keywords: ischemic; preconditioning; congenital heart disease
MeSH Terms: conditions — Heart Defects, Congenital; Ischemia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preconditioning (Experimental): Children who received the preconditioning stimulus
  Interventions: Procedure: Remote ischemic preconditioning
- Control (No Intervention): Children who did not receive the preconditioning stimulus

INTERVENTIONS:
Procedure: Remote ischemic preconditioning — Remote ischemic preconditioning was induced by four 5-minutes cycles of lower limb ischemia and reperfusion using a blood pressure cuff
  Other Names: Inicial letters of the full name; Register number provided by hospital
  Arms: Preconditioning

SUMMARY:
The study research is to analyse brief episodes of limb ischemia applied to children the day before open heart surgery as protection from myocardial injury induced by extracorporeal circulation.

DETAILED DESCRIPTION:
Children undergoing repair of congenital heart defects were randomized to RIPC (remote ischemic preconditioning) or control treatment. RIPC was induced by four 5-minutes cycles of lower limb ischemia and reperfusion using a blood pressure cuff. Measurements of troponin I, brain natriuretic peptide, interleukines 8 and 10, real time PCR to NFKB and clinical parameters were obtained and compared postoperatively (4, 12, 24 and 48 hous after).

ELIGIBILITY:
Inclusion Criteria:

* 1 month to 2 years age
* waiting for open heart surgery in hospital
* 2008, january to march
* Rachs-1, except the 1 category

Exclusion Criteria:

* genetic syndromes
* infected children
* immunodeficiency
* immunosuppressor use
* no parents permission

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2008-01; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula CP Carlotti, 1, Study Director — University of Sao Paulo
Locations (1):
- General Hospital of Ribeirao Preto, Sao Paulo University, Ribeirão Preto, São Paulo, Brazil

RESULTS

PARTICIPANT FLOW:
Groups:
- Preconditioning: Children who received the preconditioning stimulus:submitted to four periods of five minutes of lower limb ischemia by using a blood pressure cuff intercalated with periods of five minutes of reperfusion, the day prior to cardiac surgery. We used the patient sistolic blood pressure plus 15 mmHg to promote de preconditioning stimulus.
Period: Overall Study
Arm/Group | Preconditioning | Control
Started | 12 | 10
Completed | 12 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Preconditioning | Control | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 12 | 10 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.9 (6.6) | 6.6 (4.6) | 7.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 7 | 6 | 13
Region of Enrollment [Number; unit: participants]
  Brazil | 12 | 10 | 22

OUTCOME MEASURES:

1. Secondary Outcome: NT-proBNP
Description: Plasma concentration of the amino-terminal of B-type natriuretic peptite (NT-proBNP)was measured by enzyme electrochemiluminescence immunoassay.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Preconditioning | Control
Number analyzed (Participants) | 12 | 10
pg/mL | 8.565 (5.155) | 12.681 (5.822)

2. Primary Outcome: IkB-alpha Expression
Description: Expressure of gene of an inhibitory protein called kappa-B alpha (IkB-alpha). Inhibits the inflammatory response protein called kappa-B nuclear factor. To measure that expression we used a real time protein chain reaction (RT-PCR), always comparing with an endogenous protein expression (this way, the encountered value is apresented in "arbitraries units", that means how much times the expression of the protein IkB-alpha is bigger than the endogenous protein that present a invariable value.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Preconditioning | Control
Number analyzed (Participants) | 12 | 10
units on a scale | 4.1 (3.7) | 3.6 (1.7)

3. Primary Outcome: Interleucine 8
Description: Quantification of interlecine 8 (a pro-inflammatory protein) using the ELISA method
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Control: Children that don´t received the preconditioning stimmulus
Arm/Group | Preconditioning | Control
Number analyzed (Participants) | 12 | 10
pg/mL | 20.8 (17.2) | 32.2 (19.4)

4. Secondary Outcome: Troponin I
Description: Seric concentration of troponin I, a myocardial cell injury marker. We measured by solid-phase chemiluminescence immunoassay.
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Preconditioning | Control
Number analyzed (Participants) | 12 | 10
pg/mL | 33.7 (21.5) | 22.3 (19.3)

ADVERSE EVENTS:
Time Frame: 1 month
Description: We searched for adverse events secondary to preconditioning in the leg, such ischemic lesions, nerve palsy or thrombus
Arm/Group | Preconditioning | Control
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 0/12 | 0/10

LIMITATIONS AND CAVEATS:
Small number of subjects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less